CLINICAL TRIAL: NCT04709861
Title: Early 2 Weeks Versus Delayed 6 Weeks Post-Operative Weight-Bearing in Total Ankle Replacement
Brief Title: TAR 2 Weeks vs 6 Weeks Post-Operative Weight-Bearing
Acronym: TAR
Status: Terminated | Type: Observational
Why Stopped: PI left the institution before enrollment was completed
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 12704
Record Dates: First submitted 2020-12-18; First posted 2021-01-14 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Ankle Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective 6 week Weight-Bearing: Delayed weight-bearing 6 weeks after total ankle replacement
- Prospective 2 week Weight-Bearing: Early weight-bearing 2 weeks after total ankle replacement

SUMMARY:
The Investigators hypothesize that an early 2 week post-operative protocol will have no difference in the successful osseointegration and stability of the total ankle replacement as compared to a delayed 6 week post-operative protocol. The importance of the research is to allow patients who receive a total ankle replacement to bear weight 4 weeks earlier than the current protocol with no negative effect on the osseointegration and stability of the ankle replacement.

DETAILED DESCRIPTION:
The study will be conducted using two groups. The first group will be a retrospective review of charts of 35 patients who received a total ankle replacement porous prosthesis by an orthopedic surgeon at the University of Oklahoma Health Sciences Center. This group was received a delayed 6 week post-operative weight-bearing protocol.

The second group will be prospective and include patients who will receive the same total ankle replacement porous prosthesis but will be assigned to early 2 weeks post-operative weight-bearing protocol.The retrospective and prospective groups will be age and gender matched. A Wright Medical Infinity Total Ankle Replacement System will be used for both groups.

Both groups will be assessed at 1 year and 2 years post-operative. This assessment will take place during the post-operative care period and will be conducted as part of their post-operative care by the operating physician.

ELIGIBILITY:
Retrospective/Prospective Inclusion Criteria:

Patients who have had a total ankle replacement with the Principal Investigator from the initiation of his clinical practice from September 2015 to September 2020.

Had delayed weight-bearing. Patients whose age and gender match the retrospective delayed weight-bearing group.

Retrospective/Prospective Exclusion Criteria:

Patients who have had Total Ankle Replacement with subsequent development of suture wound infection.

Patients who have had Total Ankle Replacement with subsequent development of deep infection requiring revision.

Patient who have had Total Ankle Replacement with subsequent development of Peri-prosthetic fractures during surgery or post-op.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 35
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
osseointegration | time of surgery through 2 years
  a Chi Square Test will take place during the post-operative care period and will be conducted as part of their post-operative care by the operating physician.

SECONDARY OUTCOMES:
stability of implant | time of surgery through 2 years
  radiological images assessment will take place during the post-operative care period and will be conducted as part of their post-operative care by the operating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Amgaad Haleem, MD, Principal Investigator — University of Oklahoma, Orthopedic Surgery
Locations (1):
- OUPhysicians, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Information will only be shared with the our own research team